CLINICAL TRIAL: NCT03757013
Title: Real Life Data for Otezla Evidence: Assessing Benefits of Apremilast in Patients With Moderate to Severe Chronic Plaque Psoriasis Followed by Dermatologists Under Real Life Settings in France
Brief Title: A Study to Assess Benefits of Apremilast in Patients With Moderate to Severe Chronic Plaque Psoriasis Followed by Dermatologists Under Real Life Settings in France
Acronym: REALIZE
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-021; U1111-1218-9791 (Registry Identifier: WHO)
Record Dates: First submitted 2018-09-25; First posted 2018-11-28 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis; Apremilast; France; CC-10004
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with Apremilast: Patients with moderate to severe chronic plaque psoriasis after failure or contra-indication or intolerance to other systemic therapy including ciclosporin, methotrexate, or phototherapy UVA + psoralen (PUVA therapy).
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast

SUMMARY:
REALIZE study will include a representative sample of 500 patients with moderate to severe plaque psoriasis for whom the treating dermatologist has decided to begin apremilast treatment in accordance with the local label reimbursement criteria. Patients may be enrolled into the study up to 4 weeks after starting the study treatment.

REALIZE is a longitudinal, multicenter, observational study under real life settings in patients with moderate to severe chronic plaque psoriasis after failure or contra-indication or intolerance to other systemic therapy including ciclosporin, methotrexate, or phototherapy UVA + psoralen (PUVA therapy).

DETAILED DESCRIPTION:
Eligible patients will be identified and invited to enroll from approximately 100 dermatologists in France practicing in public hospitals (or private clinics) or private practice. Patients will be followed over 12 months after initiation of apremilast or until discontinuation of apremilast whatever the earlier. Given the observational nature of the study, apremilast dosing and duration will be at the sole discretion of the treating dermatologist, in accordance with the local label and daily clinical practice. Patient care will follow routine clinical practice, involving regular follow-up visits, without any mandatory visit. In daily practice, patients are usually seen by their treating dermatologist every 6 months. In this study, patients will be followed up at most 12 months after apremilast initiation.

During this study, it is expected to collect data at inclusion (enrolment visit) and around 6 months and 12 months after apremilast initiation, on electronic case report forms (eCRF) by the dermatologist after performing a visit around 6 and 12 months to evaluate the treatment response following the apremilast initiation.

Due to the observational nature of the study, the study protocol does not require any specific tests or additional examinations. All assessments will be recorded in the electronic case report form (eCRF) according to the normal practice of the treating dermatologist. Self-questionnaires will be filled by the patient when visiting his/her dermatologist.

Total duration of the study is 2 years and 6 months, which includes an enrollment period of 1 year and 6 months and a follow up period of up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged at least 18 years
* Patient with a diagnosis of stable moderate to severe chronic plaque psoriasis
* For whom the treating dermatologist has made the decision to initiate apremilast treatment in accordance with the local label and reimbursement criteria i.e. a history of failure or contra-indication or intolerance to other systemic therapy including ciclosporin, methotrexate, or phototherapy UVA + psoralen (PUVA therapy)
* Patient having started apremilast up to 4 weeks before the enrolment visit for treatment of moderate to severe chronic plaque psoriasis even if apremilast has been stopped before inclusion in the study
* Patient literate and willing to fill in questionnaires
* Non-opposition form signed by the investigator indicating that the patient received information about the study, and orally agreed.

Exclusion Criteria:

* Patient who refuses to participate in the study or is unable to give his/her oral consent
* Patient having participated in an interventional study in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe plaque psoriasis for whom the treating dermatologist has decided to begin apremilast treatment in accordance with the local label reimbursement criteria. Patients may be enrolled into the study up to 4 weeks after starting the study treatment.
  All eligible patients will be included in the safety population in consecutive order based on the date of the non-opposition form.
  However, only patients who have completed 6 (± 1) months of treatment will be included in the reference analysis population
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Patient Benefit Index score (PBI-S) ≥1 at 6 months after initiation of apremilast. | Up to 6 months
  The PBI-S questionnaire for skin diseases is a validated instrument to assess treatment needs and benefits in patients with skin diseases. It comprises 23 items on patient-relevant therapy needs and benefits.

SECONDARY OUTCOMES:
Proportion of subjects with PBI-S (range 0-4) at 6 months after apremilast initiation | Up to 6 months
  The PBI-S questionnaire for skin diseases is a validated instrument to assess treatment needs and benefits in patients with skin diseases. It comprises 23 items on patient-relevant therapy needs and benefits.
Proportion of patients with PBI-S=4 at 6 months after apremilast initiation | Up to 6 months
  The PBI-S questionnaire for skin diseases is a validated instrument to assess treatment needs and benefits in patients with skin diseases. It comprises 23 items on patient-relevant therapy needs and benefits
Adherence Rate | Up to 12 months
  The adherence rate will be defined as the percentage of patients pursuing the treatment with apremilast at 12 months after the initiation of apremilast.. The calculation will take into account the patients having started and discontinued apremilast within 4 weeks before the enrolment visit.
Percentage of patients substituting apremilast | Up to 24 months
  The percentage of patients substituting apremilast by a biologic will be estimated by the Kaplan Meier method. The date of origin will be defined as the date apremilast has been started.
Dermatology Life Quality Index (DLQI) | Up to 24 months
  DLQ is a 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument. It covers a variety of health dimensions, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period is 7 days. Each item is graded on a Likert scale of 0-3, which gives an overall score ranging from 0 to 30 where lower scores mean better quality of life.
Proportion of patients with DLQI ≤ 5 | Up to 24 months
  DLQ is a 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument. It covers a variety of health dimensions, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period is 7 days. Each item is graded on a Likert scale of 0-3, which gives an overall score ranging from 0 to 30 where lower scores mean better quality of life.
Proportion of patients achieving DLQI 0/1 | Up to 24 months
  DLQ is a 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument. It covers a variety of health dimensions, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period is 7 days. Each item is graded on a Likert scale of 0-3, which gives an overall score ranging from 0 to 30 where lower scores mean better quality of life.
Change in DLQI score from M0 to M6 and M12 | Up to 12 months
  DLQ is a 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument. It covers a variety of health dimensions, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period is 7 days. Each item is graded on a Likert scale of 0-3, which gives an overall score ranging from 0 to 30 where lower scores mean better quality of life.
Proportion of patients with improvement in DLQI ≥ 5 points between M0 and M6, M12 | Up to 12 months
  DLQ is a 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument. It covers a variety of health dimensions, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period is 7 days. Each item is graded on a Likert scale of 0-3, which gives an overall score ranging from 0 to 30 where lower scores mean better quality of life.
Treatment Satisfaction Questionnaire for Medication (TSQM9) | Up to 24 months
  TSQM-9 is a 9-item validated self-administered questionnaire used to evaluate the patient's overall satisfaction with study treatment. The TSQM-9 consists of 8 items that make up 3 specific scales (effectiveness, side effects, convenience) and one global satisfaction scale. Scale scores are transformed into scores from 0 to 100 with higher scores representing higher satisfaction in that domain.
Proportion of patients with sPGA 0 or 1 | Up to 24 months
  sPGA static physician global assessment is defined as single-item-5-point categorized scale reflecting the physician's assessment of psoriasis severity. This scale ranges from 0 to 4.
Change in sPGA from baseline to M6 and M12 | Up to 12 months
  sPGA static physician global assessment is defined as single-item-5-point categorized scale reflecting the physician's assessment of psoriasis severity. This scale ranges from 0 to 4.
Percentage of BSA (%BSA) involved at M0, M6, M12 | Up to 12 months
  BSA is the measurement of the body area involved in relation to the whole body surface
Change in % BSA from M0 to M6, M12 | Up to 12 months
  BSA is the measurement of the body area involved in relation to the whole body surface
Psoriasis Area Severity Index (PASI) at M0, M6, M12 | Up to 12 months
  PASI is a common clinical tool used to measure the severity and extent of psoriasis. PASI score is a composite score grading the severity of psoriasis in four body regions according to erythema, scaling, and thickness, and the total area of skin affected. The final composite score ranges from 0 to 72, with a higher score indicating a greater severity of psoriasis
Change in PASI from M0 to M6, M12 | Up to 12 months
  PASI is a common clinical tool used to measure the severity and extent of psoriasis. PASI score is a composite score grading the severity of psoriasis in four body regions according to erythema, scaling, and thickness, and the total area of skin affected. The final composite score ranges from 0 to 72, with a higher score indicating a greater severity of psoriasis
Proportion of patients achieving PASI50 at M6, M12 | Up to 12 months
  PASI is a common clinical tool used to measure the severity and extent of psoriasis. PASI score is a composite score grading the severity of psoriasis in four body regions according to erythema, scaling, and thickness, and the total area of skin affected. The final composite score ranges from 0 to 72, with a higher score indicating a greater severity of psoriasis
Proportion of patients achieving PASI75 at M6, M12. | Up to 12 months
  PASI is a common clinical tool used to measure the severity and extent of psoriasis. PASI score is a composite score grading the severity of psoriasis in four body regions according to erythema, scaling, and thickness, and the total area of skin affected. The final composite score ranges from 0 to 72, with a higher score indicating a greater severity of psoriasis
Adverse Events (AEs) | Up to 24 months
  Number of participants with adverse events
Duration of disease | Baseline
  Duration of disease will be defined as the length of time the disease has been present, indication by months of years.
Number of areas of plaque psoriasis | Baseline
  The number of area of plaque psoriasis will be defined by the number of area observed by the Investigator
Type of chronic psoriasis involved | Baseline
  Types if chronic psoriasis, scalp, palmoplantar, genital
The number of lines of previous systemic treatments | Baseline
  Number of lines of previous systemic treatments will be described by one line, two lines
Type of systemic therapy previously administered | Baseline
  The type of systemic therapies includes corticosteroids, topical, other classification of medications
Duration of previous chronic psoriasis treatment | Baseline
  The duration of previous treatment will be described in months, years.
Number of motivations of the prescription of apremilast | Up to 24 months
  Motivations will be described by the number of patients with lack of response or intolerance or patient's dissatisfaction regarding the previous treatment.
Percentage of motivations of the prescription of apremilast | Up to 24 months
  Motivations will be described by the percentage of patients with lack of response or intolerance or patient's dissatisfaction regarding the previous treatment.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (93):
- France (93):
  - Private Practice, Amiens, Amiens
  - Saint-Joseph Clinic, Angouleme, Angoulême
  - Private Practice, Antibes, Antibes
  - Private Practice 2, Antony, Antony
  - Private Practice 2, Arcachon, Arcachon
  - Private Practice, Argenteuil, Argenteuil
  - Private Practice, Aubière, Aubière
  - Private Practice, Auch, Auch
  - Auxerre Hospital, Auxerre
  - Henri Duffaut Hospital, Avignon
  - Private Practice, Besançon, Besançon
  - Reims-Bezannes Polyclinic 2, Bezannes
  - Reims-Bezannes Polyclinic 3, Bezannes
  - Reims-Bezannes Polyclinic, Bezannes
  - Private Practice, Bègles, Bègles
  - Private Practice, Biarritz, Biarritz
  - Private Practice, Bordeaux, Bordeaux
  - Docteur Duchenne Hospital 2, Boulogne-sur-Mer
  - Docteur Duchenne Hospital, Boulogne-sur-Mer
  - Private Practice 2, Caen, Caen
  - Private Practice 3, Caen, Caen
  - Private Practice, Caen, Caen
  - Private Practice, Cannes, Cannes
  - Private Practice, Chamalières, Chamalières
  - Métropole Savoie Hospital, Chambéry
  - Trousseau Hospital, Chambray-lès-Tours
  - Private Practice 2, Chartres, Chartres
  - Private Practice, Chartres, Chartres
  - Private Practice 2, Chalons-en-Champagne, Châlons-en-Champagne
  - Private Practice, Chalons-en-Champagne, Châlons-en-Champagne
  - Chalons-en-Champagne Hospital, Châlons-en-Champagne
  - New Sud Francilien Hospital, Corbeil-Essonnes
  - GH de Dax, Dax, Dax
  - Private Practice 2, Dijon, Dijon
  - Private Practice 3, Dijon, Dijon
  - Private Practice, Dijon, Dijon
  - Private Practice, Dole, Dole
  - Victor Jousselin Hospital, Dreux
  - Private Practice, Essey-les-Nancy, Essey-lès-Nancy
  - Emile Durkheim Hospital - Saint Jean Health Center, Épinal
  - Golfe de St-Tropez Clinic, Gassin
  - Private Practice 2, Joue les Tours, Joué-lès-Tours
  - Private Practice 3, Joue les Tours, Joué-lès-Tours
  - Private Practice, Joue les Tours, Joué-lès-Tours
  - Private Practice, L'Union, L'Union
  - Private Practice 2, La Teste-de-Buch, La Teste-de-Buch
  - Private Practice, La Teste-de-Buch, La Teste-de-Buch
  - Private Practice, La Valette du Var, La Valette-du-Var
  - Private Practice, La Varenne Saint Hilaire, La Varenne-Saint-Hilaire
  - Private Practice 2, Laval, Laval
  - Private Practice, Laval, Laval
  - Private Practice, Le-Bourget-du-Lac, Le Bourget-du-Lac
  - Private Practice, Le Mans, Le Mans
  - Mans Hospital 2, Le Mans
  - Mans Hospital, Le Mans
  - Private Practice, Lille, Lille
  - Private Practice 2, Luce, Lucé
  - Private Practice, Luce, Lucé
  - Private Practice, Lyon, Lyon
  - Edouard Herriot Hospital, Lyon
  - Private Practice 2, Lyon, Lyon
  - Private Practice 4, Lyon, Lyon
  - Private Practice, Martigues, Martigues
  - Annecy Genevois Hospital, Metz Tessy, Metz-Tessy
  - Private Practice, Meudon-la-Forêt, Meudon-la-Forêt
  - Private Practice, Muret, Muret
  - Hotel Dieu Hospital, Dermatologic Clinic, Nantes
  - Private Practice, Narbonne, Narbonne
  - Private Practice, Nevers, Nevers
  - Private Practice 2, Nice, Nice
  - Private Practice 3, Nice, Nice
  - Private Practice, Nogent-Le-Rotrou, Nogent-le-Rotrou
  - Private Practice, Orléans, Orléans
  - Private Practice, Paris, Paris
  - Private Practice 2, Paris, Paris
  - Private Practice 3, Paris, Paris
  - Private Practice 4, Paris, Paris
  - Private Practice 5, Paris, Paris
  - Private Practice, Pontarlier, Pontarlier
  - Private Practice, Pontoise, Pontoise
  - Private Practice, Quimper, Quimper
  - CHI de Cornouaille - Laennec, Quimper
  - Mathilde II Clinic, Rouen
  - Private Practice, Saint-Etienne, Saint-Etienne
  - Saint-Etienne Hospital, Saint-Priest-en-Jarez
  - Private Practice, Torcy, Torcy
  - BCRM Toulon - HIA Saint-Anne, Toulon
  - Private Practice, Toulouse, Toulouse
  - Nord Franche-Comté Hospital, Trévenans
  - Valence Hospital 2, Valence
  - Valence Hospital 3, Valence
  - Valence Hospital, Valence
  - Jacques Lacarin Hospital, Vichy

REFERENCES:
- [Derived] Jullien D, Richard MA, Halioua B, Bessette C, Derancourt C, Bouloc A. The Needs of Patients with Psoriasis and Benefits of Apremilast in French Clinical Practice: Results from the Observational REALIZE Study. Dermatol Ther (Heidelb). 2023 Jun;13(6):1361-1376. doi: 10.1007/s13555-023-00933-z. Epub 2023 May 19. PMID 37204608
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com